CLINICAL TRIAL: NCT03904433
Title: Quantification of Ketosis After Intake of Coconut Oil and Caprylic Acid-With and Without Glucose-After a 12-hour Fast: A 6-way Cross-over Study in Healthy Older Adults
Brief Title: Quantification of Ketosis After Intake of Coconut Oil and Caprylic Acid-With and Without Glucose-After a 12-hour Fast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Miia Kivipelto, Professor, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CC1
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Aged
MeSH Terms: interventions — Coconut Oil; octanoic acid; Sunflower Oil; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1. Sunflower oil (Experimental): Sunflower oil (30 g)
  Interventions: Other: Sunflower oil
- 2. Caprylic acid (Experimental): Caprylic acid (20 g) + Sunflower oil (10 g)
  Interventions: Dietary Supplement: Caprylic acid; Other: Sunflower oil
- 3. Caprylic acid + Glucose (Experimental): Caprylic acid (20 g) + Sunflower oil (10 g) + Glucose (50 g)
  Interventions: Dietary Supplement: Caprylic acid; Other: Sunflower oil; Other: Glucose
- 4. Coconut oil (Experimental): Coconut oil (30 g)
  Interventions: Other: Coconut oil
- 5. Coconut oil + Glucose (Experimental): Coconut oil (30 g) + Glucose (50 g)
  Interventions: Other: Coconut oil; Other: Glucose
- 6. Coconut oil + Caprylic acid (Experimental): Coconut oil (30 g) + Caprylic acid (20 g)
  Interventions: Other: Coconut oil; Dietary Supplement: Caprylic acid

INTERVENTIONS:
Other: Coconut oil — Coconut oil given in coffee with cream
  Arms: 4. Coconut oil; 5. Coconut oil + Glucose; 6. Coconut oil + Caprylic acid
Dietary Supplement: Caprylic acid — Caprylic acid given in coffee with cream
  Arms: 2. Caprylic acid; 3. Caprylic acid + Glucose; 6. Coconut oil + Caprylic acid
Other: Sunflower oil — Sunflower oil given in coffee with cream
  Arms: 1. Sunflower oil; 2. Caprylic acid; 3. Caprylic acid + Glucose
Other: Glucose — Glucose dissolved in water
  Arms: 3. Caprylic acid + Glucose; 5. Coconut oil + Glucose

SUMMARY:
In a cross-over design, 15 participants, age 65-75, will be tested in six different arms in a randomised order. After a 12-hour fast participants will be served 2.5 dl coffee with 15 g cream + 30-50 g of different fatty acids, with or without 50 g glucose. Blood ketones and other biomarkers will be measured during 4 hours.

DETAILED DESCRIPTION:
In the metabolic state ketosis, beta-hydroxybutyrate (BHB) and acetoacetate are synthesised from fatty acids in the liver, resulting in higher circulating levels. Ketosis can be induced by fasting or adherence to a low-carb-high-fat diet, but also by intake of-at least some-medium-chain-triglycerides (MCT). MCT are built from fatty acids with a chain of 6-12 carbon atoms. Caprylic acid (C8) is well known to be ketogenic, but the effect of lauric acid (C12)-constituting about 50% of coconut oil-is less clear.

The aim of this study is to assess ketosis, as a combined effect of an extended overnight fast, and intake of coconut oil or C8, and to study how ketosis is affected by simultaneous glucose intake. Sunflower oil is used as control, expected to not break fasting ketosis, although not being ketogenic in itself. Some sunflower oil is also added to C8 to make that arm isocaloric with coconut oil, with a roughly similar proportion of MCT.

Coffee with cream will be used as a vehicle, and although coffee has been reported to be mildly ketogenic, this effect is expected to be negligible and equally distributed between arms.

ELIGIBILITY:
Inclusion Criteria:

* Daily consumption of coffee
* Written informed consent

Exclusion Criteria:

* Smoker
* Weight <50 kg
* Diagnosed diabetes
* History of heart disease
* History of disease related to internal organs or metabolism
* Experience of "sensitive gut", or known intolerance to the test ingredients
* Medication expected to affect glucose- or lipid-metabolism
* Fasting during study or one month before
* High intensity physical activity > 3 times/week
* Dementia
* Severe psychiatric conditions
* Hb<125 g/L
* Participation in other lifestyle intervention last 6 months

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Concentrations of BHB, area under the curve, 0-4 h | 0, 15, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240 (minutes)
  BHB, measured in venous whole blood with a point-of-care meter

SECONDARY OUTCOMES:
Concentrations of total ketones | 0, 30, 60, 120 (minutes)
  BHB + acetoacetate, laboratory analyses from plasma
Concentrations of BHB (capillary) | 30, 60, 120 (minutes)
  BHB, measured in capillary whole blood with a point-of-care meter, for exploratory comparisons. (not measured in arm 3 & 5)
Concentrations of BDNF / pro-BDNF | 0, 60, 120, 240 (minutes)
  Brain-derived neurotrophic factor (BDNF) & pro-BDNF in serum (not measured in arm 2, 3 & 5)
Concentrations of glucose | 0, 60, 120, 180, 240 (minutes)
  Glucose, laboratory analysis
Self-rated satiety | 240 (minutes)
  Assessed by a 5-grade categorical hunger-scale in a questionnaire at the end of each testing session. Participants will be instructed to choose the most suitable description of their hunger:
  1. Not hungry at all.
  2. Modestly hungry. Lunch can wait.
  3. It feels like the right time for lunch. Hunger appeared during the last hour.
  4. Very hungry. Hunger appeared during the last hour.
  5. Hungry or very hungry. Hunger has been palpable for more than one hour.
  Answers a, b & c will be interpreted as sufficient satiety.
Self-rated tolerance of beverage | 240 (minutes)
  Assessed by a 4-grade categorical scale in a questionnaire at the end of each testing session:
  Did you experience any inconvenience (i.e. nausea, upset stomach), which you attribute to the beverage you were served today?
  1. No
  2. Yes, minor inconvenience.
  3. Yes, moderate inconvenience.
  4. Yes, major inconvenience.
  If the answer is b, c or d participants are asked to give a short description.

OTHER OUTCOMES:
Concentrations of insulin | 0, 60, 90, 120, 240 (minutes)
  Not measured at minutes 60, 90 & 120 in arm 1, 2, 4, 6
Concentrations of glucagon | 0, 60, 90, 120, 240 (minutes)
  Not measured at minutes 60, 90 & 120 in arm 1, 2, 4, 6
Concentrations of HbA1c | 0 (minutes)
  Only measured at the first testing session

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Stockholm County, Sweden

REFERENCES:
- [Derived] Norgren J, Daniilidou M, Kareholt I, Sindi S, Akenine U, Nordin K, Rosenborg S, Ngandu T, Kivipelto M, Sandebring-Matton A. Serum proBDNF Is Associated With Changes in the Ketone Body beta-Hydroxybutyrate and Shows Superior Repeatability Over Mature BDNF: Secondary Outcomes From a Cross-Over Trial in Healthy Older Adults. Front Aging Neurosci. 2021 Aug 20;13:716594. doi: 10.3389/fnagi.2021.716594. eCollection 2021. PMID 34489682
- [Derived] Norgren J, Sindi S, Sandebring-Matton A, Kareholt I, Daniilidou M, Akenine U, Nordin K, Rosenborg S, Ngandu T, Kivipelto M. Ketosis After Intake of Coconut Oil and Caprylic Acid-With and Without Glucose: A Cross-Over Study in Healthy Older Adults. Front Nutr. 2020 Apr 15;7:40. doi: 10.3389/fnut.2020.00040. eCollection 2020. PMID 32351966